CLINICAL TRIAL: NCT02800473
Title: Evaluation of an Innovative Medical Device Made of a Bimodal Endoscopic Imager and of a Software for Panoramic Images Building of the Bladder Inner Wall (French National Research Agency, CyPaM2 Project, ANR-11-TECS-001) (CyPaM2)
Brief Title: Validation of Endoscopic Bimodal Imager for the Bladder Cancer Detection
Acronym: CyPaM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A01297-42
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Hexvix; Bimodal Endoscopic Imager; Cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Other): Patients with a suspicion of a bladder cancer or suspected recurrence of bladder cancer will have a cystoscopy under their care.
  Patients will be randomized to know the order of carrying out cystoscopy with one or the other medical devices.
  24 hours and 48 hours after the exam, a nurse will contact the patient to detect potential adverse effects
  Interventions: Device: Strorz (commercial); Device: CyPaM2 (experimental)

INTERVENTIONS:
Device: Strorz (commercial)
Device: CyPaM2 (experimental)

SUMMARY:
This study evaluates the therapeutic value of: (i) simultaneous endoscopic visualization of the inner bladder using white light and blue light excitations and (ii) high resolution panoramic images of the bladder inner wall.

All participants will undergo fluorescence cystoscopy: the first half using first a reference medical device for fluorescence cystoscopy already on the market then using the innovative device specifically developped for the CyPaM2 project.

The other half will undergo fluorescence cystoscopy using first the innovative then the reference medical device.

DETAILED DESCRIPTION:
An innovative medical device was developped by the CyPaM2 project's partners.This device is made of a hardware and of a software part: (i) an imager (light source and sensors) for simultaneous and colocalized visualisation of the bladder using white light and blue light for fluorescence excitation and (ii) a mosaicing software for automatic building of high-resolution panoramic images of the bladder inner wall. The medical device's qualitative (human engineering, images qualitty) and quantitative (medical examination and panoramic images building durations) specifications will be evaluated during the clinical trial in comparison with a reference medical device already on the market. The main goals are to achieve (i) better sensitivity of bladder cancers' cystocopic diagnosis and shorter medical examination durations thanks to the simultaneous visualization of the bladder inner wall with white and blue lights and (ii) better patients' follow up thanks to the high resolved panoramic images.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient with suspicion of a bladder cancer or a suspected recurrence of a bladder cancer
* Cytological and bacteriological examination of urine culture negative
* Patient must be affiliated to a social security system
* Ability to provide written informed consent patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study

Exclusion Criteria:

* Age < 18 years
* Bladder infection in progress and untreated
* Hemorrhage
* Urethral stenosis
* Contraindication for a cystoscopy examination
* Contraindication to administration of Hexvix (porphyria, hypersensitivity to hexylaminolévulinate or excipient of Hexvix (disodium phosphate dihydrate, potassium dihydrogen phosphate)
* Pregnant or breast feeding females
* Patients deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Ergonomic comparaison of the two devices | 1 day
  Ergonomic of the two devices will be evaluated and compared by using the scale NASA TLX (Hart SG, et al., 1998).

SECONDARY OUTCOMES:
Comparison of performing time | 1 day
  Performing time of medical examination with both devices will be evaluated and compared
Quality assessment of image | 1 day
  Image quality : sharpness and colorimetry will be assessed by the physician using a self-questionnaire.
Quality assessment of device evaluation | 1 day
  Device quality : sensitivity and accuracy will be assessed by the urologist using a self-questionnaire
Evaluation of recording capacity of the video sequences to perform real-time image mosaics | 1 day
  Recording capacity of the video sequences to perform real-time image mosaics will be assessed by the physician using a self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: ESCHWEGE PASCAL, Pr, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amouroux M, Salleron J, Huin-Schohn C, Ali S, Berthaud S, Rizo P, Schneider S, Vever-Bizet C, Bourg-Heckly G, Guillemin F, Le Coupanec P, Galbrun E, Daouk J, Daul C, Blondel W, Eschwege P. Clinical evaluation of a device providing simultaneous white-light and fluorescence video streams as well as panoramic imaging during fluorescence assisted-transurethral resection of bladder cancer. J Opt Soc Am A Opt Image Sci Vis. 2019 Nov 1;36(11):C62-C68. doi: 10.1364/JOSAA.36.000C62. PMID 31873695